CLINICAL TRIAL: NCT02483273
Title: Alterations of Conjunctival Microcirculation in Brain Dead Patients
Status: Completed | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tomas Tamosuitis, Lithuanian University of Health Sciences Intensive Care Clinic Research Fellow, Lithuanian University of Health Sciences
Other Study IDs: P1-BE-2-19/2011
Record Dates: First submitted 2015-06-18; First posted 2015-06-26 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Brain Death
Keywords: Conjunctival microcirculation; Sublingual microcirculation; Sidestream Dark Field (SDF) microscopy
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Brain dead patients: Brain dead patients certified by cerebral angiography.
- Healthy volunteers: Any person with no known cerebral pathology.

SUMMARY:
Study hypothesize that ocular microcirculation is reflecting cerebral perfusion. The purpose of this study is to evaluate ocular microcirculation in brain dead patients using side dark field (SDF) videomicroscope and compare it with microcirculatory parameters of healthy volunteers.

DETAILED DESCRIPTION:
Microcirculation videomicroscopy techniques are used to evaluate a global organ perfusion in various critical conditions using limited suitable sites available for visualisation. However, ocular microcirculation may become a window to specifically cerebral perfusion due to related blood supply, close anatomical proximity and easy accessibility for videomicroscopy. Cerebral perfusion mainly depends on cerebral flow and intracranial pressure and therefore we aim, for the first time, to demonstrate microcirculatory status of ocular conjunctiva in clinical conditions when cerebral flow is completely absent.

In a single center open label observational study investigators analyzed conjunctival and sublingual microcirculation using SDF videomicroscopy in brain dead patients after reaching systemic hemodynamic targets to optimise perfusion of donor organs. All brain death diagnoses were confirmed by cerebral angiography. Microcirculatory images obtained and analyzed using standardized published recommendations by experts in this field. Microcirculation of sublingual and conjunctival areas were recorded in matching number of healthy volunteers using same techniques.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed brain dead

Exclusion Criteria:

* Conjunctival or sublingual mucosa damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All single center tertiary level Neurosurgery Intensive Care unit patients angiographically confirmed brain dead.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-05; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Microvascular flow index (MFI) of ocular conjunctiva. | After confirmed diagnosis of brain death of any course using cerebral angiography at any time up to 24 hours.
  Conjunctival convective oxygen transport presented as MFI of small vessels mostly capillaries with diameter cutoff value of 20µm. Images of microcirculation were taken from at least three different points in each ocular conjunctiva and recorded for at least 20 seconds avoiding pressure artifacts. Microcirculation images were obtained using SDF videomicroscopy (Microscan®, Microvision Medicals, Amsterdam, Netherlands). Data recorded to the hard drive of personal computer using AVA 3.0v software (Microvision Medical, Amsterdam, Netherlands). Video clips were then randomly blinded and later analyzed by 2 independent investigators.
Total vessel density (TVD) of ocular concunctiva. | After confirmed diagnosis of brain death of any course using cerebral angiography at any time up to 24 hours.
  Conjunctival microvascular diffusion distance presented as TVD (mm/mm²) of small vessels mostly capillaries with diameter cutoff value of 20µm. Images of microcirculation were taken from at least three different points in each ocular conjunctiva and recorded for at least 20 seconds avoiding pressure artifacts. Microcirculation images were obtained using SDF videomicroscopy (Microscan®, Microvision Medicals, Amsterdam, Netherlands). Data recorded to the hard drive of personal computer using AVA 3.0v software (Microvision Medical, Amsterdam, Netherlands). Video clips were then randomly blinded and later analyzed by 2 independent investigators.
Perfused vessel density (PVD) of ocular conjunctiva. | After confirmed diagnosis of brain death of any course using cerebral angiography at any time up to 24 hours.
  Conjunctival microvascular diffusion distance presented as PVD (mm/mm²) of small vessels mostly capillaries with diameter cutoff value of 20µm. Images of microcirculation were taken from at least three different points in each ocular conjunctiva and recorded for at least 20 seconds avoiding pressure artifacts. Microcirculation images were obtained using SDF videomicroscopy (Microscan®, Microvision Medicals, Amsterdam, Netherlands). Data recorded to the hard drive of personal computer using AVA 3.0v software (Microvision Medical, Amsterdam, Netherlands). Video clips were then randomly blinded and later analyzed by 2 independent investigators

SECONDARY OUTCOMES:
Microvascular flow index (MFI) of sublingual mucosa. | After confirmed diagnosis of brain death of any course using cerebral angiography at any time up to 24 hours.
  Sublingual mucosa convective oxygen transport presented as MFI of small vessels mostly capillaries with diameter cutoff value of 20µm. Images of microcirculation were taken from at least three different points in sublingual mucosa and recorded for at least 20 seconds avoiding pressure artifacts. Microcirculation images were obtained using SDF videomicroscopy (Microscan®, Microvision Medicals, Amsterdam, Netherlands). Data recorded to the hard drive of personal computer using AVA 3.0v software (Microvision Medical, Amsterdam, Netherlands). Video clips were then randomly blinded and later analyzed by 2 independent investigators.
Total vessel density (TVD) of sublingual mucosa. | After confirmed diagnosis of brain death of any course using cerebral angiography at any time up to 24 hours.
  Sublingual mucosa microvascular diffusion distance presented as TVD (mm/mm²) of small vessels mostly capillaries with diameter cutoff value of 20µm. Images of microcirculation were taken from at least three different points in sublingual mucosa and recorded for at least 20 seconds avoiding pressure artifacts. Microcirculation images were obtained using SDF videomicroscopy (Microscan®, Microvision Medicals, Amsterdam, Netherlands). Data recorded to the hard drive of personal computer using AVA 3.0v software (Microvision Medical, Amsterdam, Netherlands). Video clips were then randomly blinded and later analyzed by 2 independent investigators.
Perfused vessel density (PVD) of sublingual mucosa. | After confirmed diagnosis of brain death of any course using cerebral angiography at any time up to 24 hours.
  Sublingual mucosa microvascular diffusion distance presented as PVD (mm/mm²) of small vessels mostly capillaries with diameter cutoff value of 20µm. Images of microcirculation were taken from at least three different points in sublingual mucosa and recorded for at least 20 seconds avoiding pressure artifacts. Microcirculation images were obtained using SDF videomicroscopy (Microscan®, Microvision Medicals, Amsterdam, Netherlands). Data recorded to the hard drive of personal computer using AVA 3.0v software (Microvision Medical, Amsterdam, Netherlands). Video clips were then randomly blinded and later analyzed by 2 independent investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Vidas Pilvinis, MD,PhD, Principal Investigator — Lithuanian UHS Intensive Care Clinic
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Backer D, Hollenberg S, Boerma C, Goedhart P, Buchele G, Ospina-Tascon G, Dobbe I, Ince C. How to evaluate the microcirculation: report of a round table conference. Crit Care. 2007;11(5):R101. doi: 10.1186/cc6118. PMID 17845716
- [Background] Goedhart PT, Khalilzada M, Bezemer R, Merza J, Ince C. Sidestream Dark Field (SDF) imaging: a novel stroboscopic LED ring-based imaging modality for clinical assessment of the microcirculation. Opt Express. 2007 Nov 12;15(23):15101-14. doi: 10.1364/oe.15.015101. PMID 19550794
- [Background] De Backer D, Ospina-Tascon G, Salgado D, Favory R, Creteur J, Vincent JL. Monitoring the microcirculation in the critically ill patient: current methods and future approaches. Intensive Care Med. 2010 Nov;36(11):1813-25. doi: 10.1007/s00134-010-2005-3. Epub 2010 Aug 6. PMID 20689916
- [Background] Schaser KD, Settmacher U, Puhl G, Zhang L, Mittlmeier T, Stover JF, Vollmar B, Menger MD, Neuhaus P, Haas NP. Noninvasive analysis of conjunctival microcirculation during carotid artery surgery reveals microvascular evidence of collateral compensation and stenosis-dependent adaptation. J Vasc Surg. 2003 Apr;37(4):789-97. doi: 10.1067/mva.2003.139. PMID 12663979
- [Background] Miller MM, Chang T, Keating R, Crouch E, Sable C. Blood flow velocities are reduced in the optic nerve of children with elevated intracranial pressure. J Child Neurol. 2009 Jan;24(1):30-5. doi: 10.1177/0883073808321050. PMID 19168816
- [Background] Ragauskas A, Matijosaitis V, Zakelis R, Petrikonis K, Rastenyte D, Piper I, Daubaris G. Clinical assessment of noninvasive intracranial pressure absolute value measurement method. Neurology. 2012 May 22;78(21):1684-91. doi: 10.1212/WNL.0b013e3182574f50. Epub 2012 May 9. PMID 22573638
- [Background] Pranskunas A, Vellinga NA, Pilvinis V, Koopmans M, Boerma EC. Microcirculatory changes during open label magnesium sulphate infusion in patients with severe sepsis and septic shock. BMC Anesthesiol. 2011 Jun 14;11:12. doi: 10.1186/1471-2253-11-12. PMID 21672227
- [Derived] Tamosuitis T, Pranskunas A, Balciuniene N, Pilvinis V, Boerma EC. Conjunctival microcirculatory blood flow is altered but not abolished in brain dead patients: a prospective observational study. BMC Neurol. 2016 Jul 11;16:95. doi: 10.1186/s12883-016-0618-z. PMID 27401581